CLINICAL TRIAL: NCT05282680
Title: An Integrated Trans-omics Approach to Diabetic Cardio-renal Complications: From Novel Discoveries to Personalized Medicine Substudy 2: The Hong Kong Diabetes Biobank
Brief Title: The Hong Kong Diabetes Biobank
Acronym: HKDB
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ronald C.W. Ma, Professor, Chinese University of Hong Kong
Other Study IDs: 2013.304; T12-402/13N (Other Grant/Funding Number: RGC Theme-based Research Scheme)
Record Dates: First submitted 2022-02-28; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes; Type 1 Diabetes; Diabetic Nephropathies; Diabetic Kidney Disease; Diabetic Angiopathies; Cardiovascular Diseases; Coronary Heart Disease; Diabetic Retinopathy; Stroke; Diabetes
Keywords: genetics; genomics; precision medicine; biomarkers; proteomics; epigenetics
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetic Nephropathies; Diabetic Angiopathies; Cardiovascular Diseases; Coronary Disease; Diabetic Retinopathy; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: Samples With DNA — The following biospecimens are collected: whole blood for extraction of DNA, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 diabetes: Subjects with a diagnosis of type 2 diabetes
- Type 1 diabetes: Subjects with a diagnosis of type 1 diabetes
- Diabetic kidney disease: Subjects with diabetic kidney disease (presence of albuminuria +/- eGFR<=60m/kg/m2) or history or presence of end stage renal disease

SUMMARY:
Asia is in the midst of an epidemic of diabetes. Epidemiological figures suggest that there are more than 110 million people affected by diabetes in China, with a significant proportion of young adults already affected. With increasingly young age of onset, the financial implications due to productivity loss and health care expenditures are colossal. As a result, prevention of diabetes and diabetic complications has been identified as a top healthcare priority in China.

In Chinese, diabetic kidney disease with albuminuria, which reflects widespread vascular damage, is a major predictor for end-stage renal failure, cardiovascular complications and death, and a major contributor to the increased healthcare burden associated with diabetes. There is an immense demand for effective tools which can accurately predict diabetes and diabetic complications.

Only few genetic factors have been consistently shown to be associated with diabetic kidney disease or other diabetic complications. Identification of genetic factors or other biomarkers predicting these complications can facilitate early identification of high risk subjects for treatment, as well as provide novel targets for drug treatment. To address this, the investigators plan to utilize both hypothesis-generating whole-genome approach as well as candidate gene-based studies to identify novel genetic, epigenetic factors as well as other biomarkers associated with the development of diabetic cardiovascular and renal complications, as well as other diabetes-related outcomes.

The Hong Kong Diabetes Biobank (HKDB) is being established in order to serve as a territory-wide diabetes register and biobank for epidemiological analyses, as well as large-scale discovery and replication of genetic and epigenetic markers, and other biomarkers relating to diabetes, diabetes complications or related outcomes. Subjects will be recruited from diabetes centres across Hong Kong, and will have detailed clinical information collected at the time of written consent and blood taking. Subjects will have detailed assessment of baseline diabetes complications through a structured clinical assessment, and will be prospectively followed up for development of different diabetes-related endpoints, as well as collection of clinical information and causes of hospitalization, along with information on medications and prescription records. This multi-centre cohort and biobank aims to improve our understanding of the epidemiology of diabetes and diabetes complications and related outcomes, as well as provide a unique resource for large-scale biomarker research to advance diabetes care and precision medicine in diabetes.

DETAILED DESCRIPTION:
The Hong Kong Diabetes Biobank leverages on the existing infrastructure of clinical assessment for people with diabetes.

Subjects undergoing routine diabetes complications screen at different diabetes centres across Hong Kong will be invited for recruitment into the Hong Kong Diabetes Biobank. Subjects will receive detailed information and explanation of the study, and written informed consent will be obtained from each subject interested in participating in the study.

As part of the routine diabetes complications assessment, all subjects will undergo a structured assessment based on the same protocol, including collection of background clinical information including demographics, diabetes duration, family history, medications and other relevant medical information. Anthropometric measurements including body weight, height, BMI will be collected. Clinical assessment include blood pressure, as well as fundus photography for assessment of diabetic retinopathy, and examination of peripheral pulses for peripheral vascular disease. Urine microalbumin will be measured using spot urine albumin/creatinine ratio. Other biochemical assessment include renal function, liver function, estimated GFR, fasting lipid profile, fasting glucose and HbA1c.

An additional 20ml blood will be obtained from each participating patient for extraction of genomic DNA, storage of serum, plasma, and for subsequent biomarker studies. Samples will be transported and processed for secure centralized storage at -80°C in dedicated facilities fitted with alarms. Samples will be identified by a unique assigned sample code. Selection and use of the samples for replication studies will be governed by the Steering Committee.

All recruited subjects will be prospectively followed up for development of diabetes complications and other clinical endpoints. Other clinical information and prescription records would be obtained from the electronic medical records.

Initial analyses would include identification of biomarkers associated with cardio-renal complications in diabetes. Subjects from the registry who have developed renal complications (diabetic kidney disease (DKD) defined as stage 3 chronic kidney disease or worse i.e. eGFR ≤60ml/min/1.73m2 and/or micro/macroalbuminuria) on prospective follow-up, will be compared to subjects free of kidney complications.

Subjects who developed cardiovascular complications (defined as new-onset acute coronary events, coronary revascularization, stroke and congestive cardiac failure) will be identified for a case: control analysis to replicate genetic predictors and other biomarkers associated with development of cardiovascular complications. Control subjects will be identified as subjects with type 2 diabetes who are free of cardiovascular events described above despite long duration of disease.

Other clinical outcomes of interest include diabetes progression and need for treatment intensification (including initiation of insulin treatment), as well as other clinical events.

ELIGIBILITY:
Inclusion Criteria:

* subjects with known diabetes

Exclusion Criteria:

* subjects not capable of giving written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with known diabetes undergoing routine diabetes complications assessment at one of the designated and participating diabetes centres in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 48000 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2063-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetic kidney disease | 1-99 years
  Diabetic kidney disease will be defined as: eGFR <60 ml/min per 1.73 m2. +/- presence of elevated urine microalbumin
  Other hospital discharge diagnoses based on eGFR or ICD-9 codes or other equivalent will be used.
  Kidney failure/end stage renal disease (ESRD) will be defined by the presence of a dialysis code (procedure codes 39.95 or 54.98), a code of kidney transplant (procedure code 55.6 or diagnosis codes 996.81 or V42.0), or eGFR <15 ml/min per1.73 m2. The onset time will be defined as the period from baseline visit to the date of kidney failure onset or the censored date, whichever came first.
  The rate of decline in eGFR and % drop in eGFR, as well as changes in urine albuminuria will also be explored as additional clinical endpoints in diabetic kidney disease.
  Identification of genetic variants or other biomarkers associated with diabetic kidney disease by association analyses may utilize one or more of the clinical definitions of diabetic kidney disease.
Cardiovascular complications in diabetes | 1-99 years
  Cardiovascular complications in diabetes will be defined as coronary heart disease (CHD), stroke, and/or peripheral vascular disease (PVD), and/or congestive heart failure.
  Coronary Heart Disease is defined as myocardial infarction, ischemic heart disease, or cardiac revascularisation.
  Stroke is defined as ischemic stroke except transient ischemic attack, hemorrhagic stroke, or acute but ill-defined cerebrovascular disease
  Peripheral vascular disease is defined as amputation, gangrene, or peripheral revascularization.
  Hospitalization for heart failure is defined as hospitalization for congestive heart failure.
  Identification of genetic variants or other biomarkers associated with cardiovascular disease in diabetes may utilize one or more of the clinical definitions of cardiovascular complications in diabetes.

SECONDARY OUTCOMES:
Diabetes progression | 1-99 years
  Diabetes glycaemic progression will be defined as:
  1. progression to continuous insulin treatment (more than 6-months' duration), or
  2. failure of non-insulin diabetes treatment (two consecutive HbA1c ≥ target, more than 3-months apart during treatment with ≥2 non-insulin diabetes therapies.
  Identification of genetic variants or other biomarkers associated with diabetes progression may utilize one or more of the above definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Ma, FRCP, Principal Investigator — Department of Medicine and Therapeutics, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for Hong Kong Diabetes Biobank — https://www.hongkongdiabetesbiobank.org/projects.aspx?id=3